CLINICAL TRIAL: NCT03207529
Title: Phase Ib Study of BYL719 (Alpelisib) in Combination With Androgen Receptor Inhibitor (Enzalutamide) in Patients With Androgen Receptor (AR)-Positive and PTEN Positive Metastatic Breast Cancer
Brief Title: Alpelisib and Enzalutamide in Treating Patients With Androgen Receptor and PTEN Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0538; NCI-2018-01127 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0538 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Advanced Breast Carcinoma; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Androgen Receptor Positive; HER2/Neu Negative; Metastatic Breast Carcinoma; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; PTEN Positive; Recurrent Breast Carcinoma; Refractory Breast Carcinoma; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Alpelisib; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (alpelisib, enzalutamide) (Experimental): Patients receive alpelisib PO and enzalutamide PO on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alpelisib; Drug: Enzalutamide

INTERVENTIONS:
Drug: Alpelisib — Given PO
  Other Names: BYL719; Phosphoinositide 3-kinase Inhibitor BYL719; Piqray
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi

SUMMARY:
This phase I trial studies the side effects and best dose of alpelisib when given together with enzalutamide in treating patients with androgen receptor and PTEN positive breast cancer that has spread to other places in the body. Alpelisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Androgen receptor can cause the growth of breast cancer cells. Hormone therapy using enzalutamide may fight breast cancer by lowering the amount of androgen the body makes. Giving alpelisib and enzalutamide may work better in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) of the combination of alpelisib (BYL719) and enzalutamide in patients with androgen receptor (AR)-positive and PTEN-positive metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To determine the dose-limiting toxicity (DLT) of the combination of BYL179 and enzalutamide.

II. To determine the safety profile of BYL179 and enzalutamide used in combination.

III. Progression-free survival (PFS) and clinical benefit rate (CBR) (complete response or partial response + prolonged stable disease) after a 16-week treatment of BYL719 and enzalutamide per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

EXPLORATORY OBJECTIVES:

I. To determine the association between aberrant circulating tumor cells (CTCs), circulating tumor deoxyribonucleic acid (ctDNA), and CBR at 16 weeks.

II. To determine the association between PIK3CA and PTEN mutations and treatment response to the combination of BYL179 and enzalutamide.

III. To determine the association between PIK3CA mutation status change in ctDNA and treatment response.

IV. To determine the molecular (CTC, ctDNA) profile of tumors that become resistant to treatment in comparison with those prior to treatment.

V. To determine the association between the AR expression level measured by immunohistochemistry (IHC) staining of tumor and CBR at 16 weeks.

OUTLINE: This is a dose-escalation study of alpelisib.

Patients receive alpelisib orally (PO) and enzalutamide PO on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >/= 18 years old.
* Patient has signed the informed consent form prior to the performance of any screening procedures and is able to comply with protocol requirements.
* Patients with central nervous system (CNS) involvement unless they meet ALL of the following criteria:

  * At least 4 weeks from prior therapy completion (including radiation and/or surgery to starting the study treatment) * Clinically and radiographically stable CNS tumor at the time of screening and not receive steroids and/or an enzyme inducing anti-epileptic mediations for brain metastasis
  * Absence of leptomeningeal disease
* Patient has metastatic breast cancer that is not suitable for surgery or radiation therapy for local disease control at the time of screening.
* Patient has disease that is hormone-receptor positive (estrogen receptor [ER] and/or progesterone receptor [PR] positive [+], HER-2/neu negative [-]) or triple-negative (ER/PR/HER-2/neu -).
* Patient has an AR-positive and PTEN-positive tumor as determined by using Clinical Laboratory Improvement Amendments (CLIA) compliant assays to identify AR-positive and PTEN-positive disease (AR positivity is defined as >= 1% of nuclear staining, PTEN positivity is defined as > 0% of nuclear staining).
* Patient has an Eastern Cooperative Oncology Group performance status (ECOG PS) =< 1 that the investigator believes is stable at the time of screening.
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin >= 9.0 g/dL
* Serum creatinine =< 1.5 x upper limit of normal (ULN)
* Total serum bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN; in the event of liver metastasis, AST/ALT =< 5 ULN
* Fasting plasma glucose (FPG) =< 140 mg/dL or =< 7.8 mmol/L
* Patient is able to swallow and retain oral medication and does not have any clinically significant gastrointestinal abnormalities that may alter drug absorption, such as malabsorption syndrome or major resection of the stomach or bowels.
* For dose-escalation cohort, patient has at least 1 measurable disease as defined by RECIST criteria (Version 1.1). For dose-expansion cohort, patient has at least 1 measurable disease as defined by RECIST criteria (version 1.1) with a lesion larger than 1.5 cm that can be biopsied by core needle biopsy.
* For dose-escalation portion of study, patients must be refractory to or intolerant of existing therapies known to provide clinical benefit for their condition.
* Patient has a life expectancy of at least 3 months in the opinion of the investigator.

Exclusion Criteria:

* Patient has a known hypersensitivity to any of the excipients of BYL719 and/or enzalutamide.
* Patient has a known or suspected primary central nervous system (CNS) tumor or CNS tumor involvement or active leptomeningeal disease.
* Patient has a history of seizures or any condition that may predispose to seizures (e.g., prior cortical stroke, significant brain trauma) at any time in the past and/or a history of loss of consciousness or transient ischemic attack within 12 months of the cycle 1, day 1 visit.
* Patient has uncontrolled diabetes.
* Patient has a history of another malignancy within 2 years prior to starting study treatment, except for cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix.
* Patient has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) (version 4.03) grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy.
* Patient has had any systemic therapy within 2 weeks prior to initiating study drug.
* Patient has participated in a prior investigational study within 3 weeks prior to initiating study drug.
* Patient has completed radiotherapy within 2 weeks prior to treatment initiation.
* Patient has any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with patient's safety, provision of informed consent, or compliance with the study procedures.
* Patient has known clinically significant cardiac disease or impaired cardiac function, such as:

  * Congestive heart failure requiring treatment (New York Heart Association grade >= 2), left ventricular ejection fraction (LVEF) < 50% as determined by multigated acquisition (MUGA) scan or ECHO.
  * History or current evidence of clinically significant cardiac arrhythmias, atrial fibrillation, and/or conduction abnormality, e.g., congenital long QT syndrome, high-grade/complete arteriovenous blockage.
  * Acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass graft, coronary angioplasty, or stenting) < 3 months prior to screening.
* Patient has a QT interval adjusted by the Fridericia formula (QTcF) > 480 msec on screening electrocardiogram (ECG).
* Patient is currently receiving medication with a known risk of prolonging the QT interval or inducing torsades de pointes (TdP) and whose treatment cannot be either discontinued or switched to a different medication prior to starting treatment with the study drug.
* Patient has any prior use of PI3K inhibitors.
* Patient has any prior use of anti-androgen therapies.
* Patient is currently receiving warfarin or other Coumarin-derived anticoagulant for treatment, prophylaxis, or other reasons. Therapy with heparin, low molecular weight heparin, or fondaparinux is allowed.
* Patient is currently receiving treatment with drugs known to be strong inhibitors or inducers of isoenzymes CYP3A or CYP2C8. The patient must have discontinued strong inducers for at least 1 week and must have discontinued strong inhibitors before the start of the study treatment. Switching to a different medication prior to initiation of the trial treatment is allowed.
* Patient has impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral BYL719 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patient has known positive serology for human immunodeficiency virus (HIV).
* Patient has any other condition that would, in the investigators' judgment, preclude the patient's participation in the clinical study due to concerns about safety or compliance with clinical study procedures; e.g., infection/inflammation, intestinal obstruction, inability to swallow oral medication, social/psychological complications.
* Patient has a history of noncompliance to medical regimens or is unable to grant consent.
* Female patients of childbearing potential have positive urine or serum pregnancy test no more than 7 days prior to starting study drug.
* Female patients of childbearing potential are not willing to use highly effective contraception to prevent pregnancy or agree to abstain from heterosexual activity throughout the study. Highly effective contraception is defined as:

  * Surgical birth control/sterilization (such as male vasectomy or female sterilization).
  * Birth control pills, injections, implants, or patches.
  * Intrauterine devices (IUDs).
  * Two barrier methods (male condom and female diaphragm, cervical cap, or sponge) in combination with a spermicide.
  * Highly effective contraception must be used by both sexes during the study and must be continued for 6 months after the last dose of study treatment. (Women of not childbearing potential: post-menopausal [age > 55 years with cessation of menses > 12 months or < 55 years but not spontaneous menses for at least 2 years or < 55 years and spontaneous menses within the past 1 year, but currently amenorrheic (e.g., spontaneous or secondary to hysterectomy), and with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone levels > 40 IU/L) or postmenopausal estradiol levels (< 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved] or who have had a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).
* Female patients who are breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of alpelisib in combination with enzalutamide | Up to 28 days

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 16 weeks
  Standard descriptive analysis will be used to summarize the data.
Profession-free survival (PFS) | Up to 16 weeks
  Will be estimated using Kaplan-Meier survival curves. From cycle 1 day 1 (cycle 1 is 28 days) to that of disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or death, whichever comes earlier, assessed up to 16 weeks]
Clinical benefit rate (CBR) (complete response or partial response + prolonged stable disease) | Up to 16 weeks
  Will be evaluated according to RECIST version 1.1. Standard descriptive analysis will be used to summarize the data.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Karuturi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org